CLINICAL TRIAL: NCT01858922
Title: Immune Reconstitution and Biomarker Identification in Patients With Newly Diagnosed Low and Intermediate Risk Hodgkins Lymphoma Receiving Chemotherapy With or Without Radiation Therapy: TXCH-HD-12A
Brief Title: Chemotherapy With or Without Radiation, Low and Intermediate Risk Hodgkins Lymphoma, TXCH-HD-12A
Acronym: TXCH-HD-12A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Carl Allen, Assistant Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-30993 TXCH-HD-12A; TXCH-HD-12A (Other: Baylor College of Medicine)
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Hodgkin Disease
Keywords: Hodgkin's Lymphoma; ABVE-PC; doxorubicin; bleomycin; vincristine; etoposide; prednisone; cyclophosphamide; DECA; decadron; cisplatin; cytarabine; Radiation
MeSH Terms: conditions — Hodgkin Disease | interventions — Doxorubicin; Bleomycin; Vincristine; Etoposide; Prednisone; Cyclophosphamide; Dexamethasone; Fumigant 93; Cytarabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rapid Early Responders (Experimental): All patients will have initial treatment utilizing ABVE-PC x2 cycles. Those patients with rapid early response (RER) determined by FDG-PET/CT scan after two cycles of ABVE-PC will receive two more cycles of ABVE-PC. If subsequent PET/CT scan indicates a complete response (CR), therapy will stop and regular follow-up will begin. If the subsequent PET/CT for RER patients indicates a partial response, those patients will undergo IFRT.
  Interventions: Drug: ABVE-PC
- Slow Early Responders (Experimental): All patients will have initial treatment utilizing ABVE-PC x2 cycles. Those patients determined to have a slow early response (SER) determined by PET/CT scan after two cycles of ABVE-PC will receive 2 courses of DECA. If after PET/CT, the patient has a partial or complete response, then 2 additional courses of ABVE-PC will be given. If subsequent PET/CT scan indicates PR or CR, those patients will then undergo IFRT.
  If stable or progressive disease is found at either PET/CT scan, the patient will be taken off-study and follow up will begin.
  Interventions: Drug: ABVE-PC; Drug: DECA

INTERVENTIONS:
Drug: ABVE-PC — Doxorubicin (A) 25mg/m2/day IV over 10min on Day 1 & Day 2
  Bleomycin (B) 5units/m2/day IV over 10min on Day 1 10units/m2/day IV over 10min on Day 8
  Vincristine (V) 1.4mg/m2/day IV push with extravasation precautions on Day 1 & 8 (Max dose 2.8mg)
  Etoposide (E) 125mg/m2/day IV over 1hr at a concentration of </=0.4mg/ml in NS on Day 1, 2 & 3
  Prednisone (P) 40mg/m2/day PO divided in 2 doses every day on Day 1-7 IV equivalent of methylprednisolone is acceptable
  Cyclophosphamide (C) 800 mg/m2 IV over 1 hr in 200 ml/m2 NS on Day 1
  Other Names: Doxorubicin (A); Bleomycin (B); Vincristine (V); Etoposide (E); Prednisone (P); Cyclophosphamide (C)
Drug: DECA — Dexamethasone (D):
  10 mg/m2 IV over 15 minutes on Day 1 and Day 2, prior to Etoposide/Cytarabine.
  Etoposide (E):
  100 mg/m2 IV over 3 hours on Day 1 and Day 2 as continuous infusion mixed with cytarabine*
  Cytarabine (A):
  3000 mg/m2 IV over 3 hours on Day 1 and Day 2 as continuous infusion mixed with etoposide*
  *Mix together in NS at an etoposide concentration of </=0.4 mg/ml
  Dexamethasone eyedrops:
  2 drops in each eye 4 times a day on Day 1, Day 2, and Day 3.
  Cisplatin (C):
  90 mg/m2 over 6 hours in 1000 ml/m2 NS + 10 gram/m2 mannitol on Day 1 as continuous infusion.
  Other Names: Dexamethasone (D); Etoposide (E); Cytarabine (A); Cisplatin (C)
  Arms: Slow Early Responders

SUMMARY:
Subjects have a type of cancer called Hodgkin Disease (HD), a cancer of the lymph system. The lymph system is made up of tissue throughout the body that makes and stores infection-fighting cells. HD is one of the most treatable childhood cancers. The standard treatment for HD involves chemotherapy (treatment with anti-cancer drugs) and radiation therapy (the use of high-dose x-rays to get rid of cancer cells). Although they are cured from their cancer, some patients experience negative side effects from treatment later in life. These kinds of side effects are often referred to as late effects. This can include problems with growth, problems with some organ functions, and sometimes second cancers. These types of effects can be associated with either chemotherapy or radiation therapy. The investigators are therefore designing studies to minimize or prevent these late effects. It is thought that if some patients can be successfully treated without radiation, those patients might experience fewer late side effects.

Some patients, however, do not respond as well to the first stages of treatment (slow early responders). Slow early responders are considered to be at higher risk for relapse. This study also looks at whether these kinds of patients will benefit from additional chemotherapy.

The purpose of this study is to look at how the immune system recovers and at how certain T-cells in the blood behave after receiving chemotherapy with or without radiation. The investigators also want to identify if bio-markers (special proteins in blood and in cancer) relate to the response of HD to study treatment.

DETAILED DESCRIPTION:
At first the subject will have 2 cycles of cancer drugs (Doxorubicin, Bleomycin, Vincristine, Etoposide, Prednisone, Cyclophosphamide). The doctors call this combination of cancer drugs ABVE-PC for short. A cycle equals 21 days. The cancer drugs will be given intravenously (IV).

Those patients evaluated as having an early response to treatment will be put in the group of Rapid Early Responders (RERs). The RER group includes those patients whose disease has been reduced by 60% or more. The next step for patients with RERs is 2 more cycles of ABVE-PC chemotherapy followed by another evaluation of their response. Those determined to have a complete response (at least an 80% disease reduction) will receive no further therapy. Those patients determined to have less than a complete response will receive radiation therapy within 6 weeks after the last cycle or when blood counts are recovered. Radiation therapy will be given to the involved areas and by the standard of care of this hospital (Texas Children's Hospital). After radiation the subject will be off treatment.

Patients with disease reduction less than 60% are put in the group of Slow Early Responders (SERs). The next step for patients with SER is 2 cycles of DECA (Dexamethasone, Etoposide, Cytarabine, and Cisplatin). On Days 1 and 2, the subject will be given dexamethasone IV first; afterwards, then they will receive the Etoposide and Cytarabine mixture. Cisplatin will be given by IV only on Day 1.

BIOLOGY TESTS The doctors are investigating molecules in tumors and blood that may help them better understand the biology of Hodgkin's Disease. These studies may also help them understand differences in patients' responses to therapy.

TISSUE FOR BIOMARKER STUDIES The doctors want to study the material that shows the make-up of the cancer (the genes of the cancer tissue) and the special "markers" of the tissue. Tissue from the subject's cancer biopsies will be used for these studies. They will collect these samples when the subject has a biopsy for clinical reasons.

IMMUNE FUNCTION AND BIOMARKER BLOOD TESTS The doctors also want to collect blood samples to study the subject's immune system and to look at biomarkers in the blood.

ELIGIBILITY:
Inclusion Criteria:

Patients with newly diagnosed, histologically confirmed Hodgkin Lymphoma (HD) who meet the following criteria:

* Stage IA and IB (non-bulky nodular lymphocyte predominant)
* Stage IIA and IIB
* Stage IIIA
* Stage IVA

Exclusion Criteria:

* Patients with Stage IA-IIA non-bulky lymphocyte predominant histology
* Patients who have received previous chemotherapy or radiation therapy (does NOT include steroids).
* Patients with symptomatic cardiac failure unrelieved by medical therapy or evidence of significant cardiac dysfunction by echocardiogram (shortening fraction <27%).
* Patients with severe renal disease (i.e. Measured or estimated creatinine clearance or radioisotope GFR <= 70 ml/min/1.73 m2).
* Patients with pre-existing severe restrictive pulmonary disease (FVC less than 60% of predicted).
* Patients with severe hepatic disease (direct bilirubin greater than 3 mg/dl or AST greater than 500 IU/L).
* Known HIV positivity
* Patients with a Karnofsky performance score <70% or Lansky score <70%.
* Female patients who are pregnant or breast feeding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-12-19 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
Response to therapy from Day 1 of Treatment | up to 18 months
  To define the general immune recovery in patients with low and intermediate risk HD undergoing chemotherapy with or without radiation therapy. Descriptive analysis of response to therapy, event-free survival, overall survival, relapse, and infection will be summarized using summary statistics.
Changes in Frequency of Regulatory Cell Population | Baseline and 3 Months
  To identify the behavior of antigen-specific cytotoxic T-cells and specific chemokine/cytokine biomarkers in patients with low and intermediate risk HD who receive chemotherapy with or without radiation therapy using means, medians, standard deviations, and confidence interval estimates. Pairwise comparisons, paired t-tests, and/or Wilcoxon signed-rank tests will be used to compare the changes.
Changes in Frequency of Regulatory Cell Population | Baseline to 6 months
  To identify the behavior of antigen-specific cytotoxic T-cells and specific chemokine/cytokine biomarkers in patients with low and intermediate risk HD undergoing chemotherapy with or without radiation therapy will be analyzed using means, medians, standard deviations, and confidence interval estimates. Pairwise comparisons, paired t-tests, and/or Wilcoxon signed-rank tests will be used to compare the changes.
Changes in Frequency of Regulatory Cell Population | Baseline to 12 Months
  To identify the behavior of antigen-specific cytotoxic T-cells and specific chemokine/cytokine biomarkers in patients with low and intermediate risk HD undergoing chemotherapy with or without radiation therapy will be analyzed using means, medians, standard deviations, and confidence interval estimates. Pairwise comparisons, paired t-tests, and/or Wilcoxon signed-rank tests will be used to compare the changes.
Changes in Frequency of Regulatory Cell Population | Baseline to 18 Months
  To identify the behavior of antigen-specific cytotoxic T-cells and specific chemokine/cytokine biomarkers in patients with low and intermediate risk HD undergoing chemotherapy with or without radiation therapy will be analyzed using means, medians, standard deviations, and confidence interval estimates. Pairwise comparisons, paired t-tests, and/or Wilcoxon signed-rank tests will be used to compare the changes.
Function of Regulatory Cell Population | Up to 18 months
  To identify tumor and circulating biomarkers in patients with low and intermediate risk HD who receive chemotherapy with or without radiation therapy and correlate with clinical outcomes including incidence of relapse and infection using random coefficient mixed models and multivariate cox proportional hazard modeling.

CONTACTS AND LOCATIONS:
Overall Officials: Carl E. Allen, MD, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States